CLINICAL TRIAL: NCT05005598
Title: Long-term Venous Catheterization in Pediatric Anesthesia: Prevalence and Risk Factors of Dysfunction.
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BOUAZIZ Hervé, Clinical Professor, Central Hospital, Nancy, France
Other Study IDs: 2021PI133
Record Dates: First submitted 2021-08-10; First posted 2021-08-13 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Catheter Dysfunction
Keywords: pediatric; thrombotic; catheter infection; mechanical complication of catheter

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pediatric population: pediatric population of CHU of Nancy, France.
  Interventions: Other: catheter dysfunction

INTERVENTIONS:
Other: catheter dysfunction — prevalence of catheter dysfunction

SUMMARY:
To evaluate the prevalence of long-life catheters dysfunction and identify the risk factors associated to premature withdrawal in pediatric population.

For that: retrospective study, during 3 years, in CHU Nancy. Data collection by informatics file after patient agreement. Primary objective: mesure prevalence of long-life catheter dysfunction

Secondary objectives:

* identify risk factors associated to premature withdrawals by thrombotic, infectious, accidental, mechanical complications.
* mesure de time spent by anethesist to put long-life catheters in emergency. Benefit of creating à vascular access unit.

ELIGIBILITY:
Inclusion Criteria:

* long-life catheter (midline, piccline, central venous catheter)
* placed in operating room
* by anesthesist
* in pédiatric population: 0 to 18 years

Exclusion Criteria:

* more than 18 years
* peripheral venous access
* not placed by anesthesist
* placed outside operating room

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric population
Sampling Method: Non-Probability Sample
Enrollment: 381 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
prevalence of premature withdrawals of long-term vascular device | Baseline (J0) is the day when the catheter is placed, up to 1 year
  the pourcentage of premature withdrawals of these catheters

SECONDARY OUTCOMES:
identify risk factors associated to premature withdrawal long-life catheter | Baseline (J0) is the day when the catheter is placed, up to 1 year
  descriptive disfunction of catheter in the medical file

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Bouaziz, PH-D, Principal Investigator — CHU NANCY
Locations (1):
- CHRU de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided